CLINICAL TRIAL: NCT06006962
Title: Aging Well Through Interactions and Scientific Education - Action Plan (AgeWISE-AP)
Acronym: AgeWISE-AP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E4828-R; I01RX004828 (NIH)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Aging
Keywords: Cognitive Aging; Lifestyle Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Two arm study: AgeWISE-AP intervention arm and a no treatment waitlist control group arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Receiving intervention - AgeWISE-AP
  Interventions: Other: Aging Well through Interactions and Scientific Education - Action Plan
- Waitlist Control (No Intervention): No intervention; will be invited to participate in intervention after completion of study.

INTERVENTIONS:
Other: Aging Well through Interactions and Scientific Education - Action Plan — 20-week program designed to provide education and individualized planning with a goal of improving brain health.
  Other Names: AgeWISE-AP
  Arms: Intervention

SUMMARY:
The purpose of this study is to learn about the effects of AgeWISE-Action Plan (AgeWISE-AP), a 20-week program designed to provide education and individualized planning with a goal of improving brain health.

DETAILED DESCRIPTION:
The overall goal of this proposal is to conduct a fully powered randomized controlled trial of a multi-component intervention designed to provide education about brain aging, improve feelings of control over brain aging, and deliver practical assistance with creation of an executable action plan (AgeWISE-Action Plan). The AgeWISE-Action Plan (AgeWISE-AP) is intended to extend our prior AgeWISE program by adding an individualized action plan component to increase older Veteran engagement in brain healthy lifestyle activities.

AIM 1 (primary): To determine whether AgeWISE-AP increases older Veterans' engagement in lifestyle factors that promote brain health. AgeWISE provides information about the differences between normal and diseased brain aging and lifestyle factors that contribute to brain health. The action plan (AP) component will use this foundation to collaboratively create an individualized brain health plan to increase Veteran engagement in brain healthy lifestyle activities. H1. AgeWISE-AP participants will demonstrate increased engagement in brain-healthy lifestyle activities compared to the control group.

AIM 2 (primary): To determine whether AgeWISE-AP improves psychological wellness. AgeWISE provides information about the relationship between cognitive aging and affective states (e.g., depression) and attitudes about aging, and teaches stress reduction techniques. The action plan (AP) will provide additional individualized supports to improve psychological well-being with personalized goals and lifestyle modifications (e.g., diet, exercise, sleep, cognitive stimulation). H2. AgeWISE-AP participants will show increases in perception of control over cognitive aging, meaning and purpose in life, quality of life, and self-efficacy, as well as improved attitudes toward aging and decreased loneliness, depression, and anxiety compared to the control group.

AIM 3 (primary): To determine whether AgeWISE-AP improves cognition. Cognitive strategies to improve cognition and functioning are presented and practiced over three AgeWISE sessions, with homework to improve generalization to day-to-day life. Engagement in brain-healthy lifestyle activities will be accomplished through the action plan (AP). H3. Self-reported memory contentment, ability, and compensatory strategy use will increase and objective cognitive testing will be better for AgeWISE-AP participants compared to the control group.

Aim 4 (exploratory): To determine whether AgeWISE-AP influences biomarkers of brain health using structural neuroimaging methods. H4. At one-year follow-up AgeWISE-AP participants will have less volumetric decline in dementia-related brain regions compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Veterans > 60 years old with concerns about brain aging who want to learn more about cognitive aging
* English speaking as all intervention materials are written in English

Exclusion Criteria:

* Veterans with impairment on a cognitive screening measure, as determined using a MoCA cutoff score for dementia of <24 OR self or other reported diagnosis of a brain disorder affecting cognition such as Alzheimer's disease, Parkinson's disease, other dementia, major stroke, or brain injury or diagnosis of psychotic disorder such as schizophrenia
* Active alcohol or substance abuse

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS) | Baseline
  Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS) is a 41-item scale that explores the frequency and duration of light, moderate, and vigorous physical activities assessed using weekly frequency and duration.
Cognitive Health Questionnaire (CHQ) | Baseline
  17-item scale that assesses frequency of various lifestyle factors, including nutritional variables and use of cognitive strategies in daily life.
Health-Promoting Lifestyle Profile II (HPLP II) | Baseline
  A 52-item questionnaire composed of six subscales including health responsibility, nutrition, physical activity, stress management, interpersonal relations, and spiritual growth. Response options are provided on a 4-point Likert scale. Subscale scores are calculated by obtaining a mean score with higher scores indicating, better outcomes.
PROMIS Social Roles and Activities | Baseline
  8 items assessing satisfaction with performing one's usual social roles and activities with response options provided on a 5-point Likert scale. A higher score represents better ability to participate or more satisfaction.
Global Sleep Assessment Questionnaire (GSAQ) | Baseline
  11 items covering mood, life activities, and medical issues as they relate to sleep and symptoms associated with disorders of sleep. Response options are provided on a 4-point Likert scale with lower scores indicating better outcomes.
General and Memory Specific Control Beliefs Scale | Baseline
  Used to measure perceived control over cognitive health. The scale is composed of two sets of items focusing on general and memory-specific control beliefs. We are interested in examining changes in memory-specific control beliefs, which include 4 items with 3 answer choices.
Philadelphia Geriatric Center Morale Scale (PGCMS) | Baseline
  17 item scale measuring dimensions of emotional adjustments in persons aged 70 to 90. It provides a multidimensional approach to assessing the state of psychological wellbeing and perceived morale using three factors: agitation, attitude toward own aging and lonely satisfaction. Total score ranges from 0-17 with higher scores indicating higher morality.
The NIH Toolbox Meaning and Purpose Short Form | Baseline
  8-item, form that assesses the degree to which participants feel their lives matter/make sense. Each item is rated on a 5-point Likert scale with responses ranging from "strongly disagree" to "strongly agree" and from "not at all" to "very much." Total score ranges from 8-40 with higher scores indicating better outcomes.
The Patient Health Questionnaire-9 (PHQ-9) | Baseline
  Reliable and valid (in a variety of patient populations) multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. Response options are provided on a 4-point Likert scale, with total score ranging from 1-27. Lower scores indicate better outcomes.
The Center for Epidemiological Studies-Depression (CES-D) | Baseline
  20-item measure that rates how often over the past week respondents have experienced depressive symptoms. Response options are provided on a 4-point Likert scale with total scores ranging from 0-60. Lower scores indicate lower depressive symptoms.
The State-Trait Anxiety Inventory (STAI) | Baseline
  Commonly used measure of anxiety with 40 total items. Response options are provided on a 4-point Likert scale. Total score range from 40-160 with lower scores indicating lower anxiety.
The General Self-Efficacy Scale (GSE) | Baseline
  10-item psychometric scale that assesses optimistic self-beliefs to cope with a variety of difficult demands in life. Response options are provided on a 4-point Likert scale with total score ranging from 10-40. Higher total score indicates better outcomes.
Multifactorial Memory Questionnaire (MMQ) | Baseline
  A measure constructed to reflect aspects of memory that are potentially amenable to clinical intervention. The Contentment subscale contains 18 statements that assess emotions and perceptions about current memory ability including anxiety, embarrassment, and irritability. The Ability subscale contains 20 items phrased as memory failures in everyday memory situations (e.g., forgetting an appointment). The Strategy subscale measures self-reported cognitive strategy use. Response options are provided on a 5-point Likert scale. Total score ranges from 0-80 with higher scores indicating better outcomes.
The Montreal Cognitive Assessment (MoCA) | Baseline
  Screening instrument that assesses multiple cognitive domains with total score ranging from 0 to 30 points, and a cut score of 24 has demonstrated very good specificity (by correctly identifying 87% of healthy participants) and excellent sensitivity when differentiating MCI (90%) and Alzheimer disease (100%) from healthy comparisons. Total score ranges from 0-30 with higher score indicating better outcomes.
Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS) | 4-months
  Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS) is a 41-item scale that explores the frequency and duration of light, moderate, and vigorous physical activities assessed using weekly frequency and duration.
Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS) | 8-months
  Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS) is a 41-item scale that explores the frequency and duration of light, moderate, and vigorous physical activities assessed using weekly frequency and duration.
Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS) | 12-months
  Community Healthy Activities Model Program for Seniors Questionnaire (CHAMPS) is a 41-item scale that explores the frequency and duration of light, moderate, and vigorous physical activities assessed using weekly frequency and duration.
Cognitive Health Questionnaire (CHQ) | 4-months
  17-item scale that assesses frequency of various lifestyle factors, including nutritional variables and use of cognitive strategies in daily life.
Cognitive Health Questionnaire (CHQ) | 8-months
  17-item scale that assesses frequency of various lifestyle factors, including nutritional variables and use of cognitive strategies in daily life.
Cognitive Health Questionnaire (CHQ) | 12-months
  17-item scale that assesses frequency of various lifestyle factors, including nutritional variables and use of cognitive strategies in daily life.
Health-Promoting Lifestyle Profile II (HPLP II) | 4-months
  A 52-item questionnaire composed of six subscales including health responsibility, nutrition, physical activity, stress management, interpersonal relations, and spiritual growth. Response options are provided on a 4-point Likert scale. Subscale scores are calculated by obtaining a mean score with higher scores indicating, better outcomes.
Health-Promoting Lifestyle Profile II (HPLP II) | 8-months
  A 52-item questionnaire composed of six subscales including health responsibility, nutrition, physical activity, stress management, interpersonal relations, and spiritual growth. Response options are provided on a 4-point Likert scale. Subscale scores are calculated by obtaining a mean score with higher scores indicating, better outcomes.
Health-Promoting Lifestyle Profile II (HPLP II) | 12-months
  A 52-item questionnaire composed of six subscales including health responsibility, nutrition, physical activity, stress management, interpersonal relations, and spiritual growth. Response options are provided on a 4-point Likert scale. Subscale scores are calculated by obtaining a mean score with higher scores indicating, better outcomes.
PROMIS Social Roles and Activities | 4-months
  8 items assessing satisfaction with performing one's usual social roles and activities with response options provided on a 5-point Likert scale. A higher score represents better ability to participate or more satisfaction.
PROMIS Social Roles and Activities | 8-months
  8 items assessing satisfaction with performing one's usual social roles and activities with response options provided on a 5-point Likert scale. A higher score represents better ability to participate or more satisfaction.
PROMIS Social Roles and Activities | 12-months
  8 items assessing satisfaction with performing one's usual social roles and activities with response options provided on a 5-point Likert scale. A higher score represents better ability to participate or more satisfaction.
Global Sleep Assessment Questionnaire (GSAQ) | 4-months
  11 items covering mood, life activities, and medical issues as they relate to sleep and symptoms associated with disorders of sleep. Response options are provided on a 4-point Likert scale with lower scores indicating better outcomes.
Global Sleep Assessment Questionnaire (GSAQ) | 8-months
  11 items covering mood, life activities, and medical issues as they relate to sleep and symptoms associated with disorders of sleep. Response options are provided on a 4-point Likert scale with lower scores indicating better outcomes.
Global Sleep Assessment Questionnaire (GSAQ) | 12-months
  11 items covering mood, life activities, and medical issues as they relate to sleep and symptoms associated with disorders of sleep. Response options are provided on a 4-point Likert scale with lower scores indicating better outcomes.
General and Memory Specific Control Beliefs Scale | 4-months
  Used to measure perceived control over cognitive health. The scale is composed of two sets of items focusing on general and memory-specific control beliefs. We are interested in examining changes in memory-specific control beliefs, which include 4 items with 3 answer choices.
General and Memory Specific Control Beliefs Scale | 8-months
  Used to measure perceived control over cognitive health. The scale is composed of two sets of items focusing on general and memory-specific control beliefs. We are interested in examining changes in memory-specific control beliefs, which include 4 items with 3 answer choices.
General and Memory Specific Control Beliefs Scale | 12-months
  Used to measure perceived control over cognitive health. The scale is composed of two sets of items focusing on general and memory-specific control beliefs. We are interested in examining changes in memory-specific control beliefs, which include 4 items with 3 answer choices.
Philadelphia Geriatric Center Morale Scale (PGCMS) | 4-months
  17 item scale measuring dimensions of emotional adjustments in persons aged 70 to 90. It provides a multidimensional approach to assessing the state of psychological wellbeing and perceived morale using three factors: agitation, attitude toward own aging and lonely satisfaction. Total score ranges from 0-17 with higher scores indicating higher morality.
Philadelphia Geriatric Center Morale Scale (PGCMS) | 8-months
  17 item scale measuring dimensions of emotional adjustments in persons aged 70 to 90. It provides a multidimensional approach to assessing the state of psychological wellbeing and perceived morale using three factors: agitation, attitude toward own aging and lonely satisfaction. Total score ranges from 0-17 with higher scores indicating higher morality.
Philadelphia Geriatric Center Morale Scale (PGCMS) | 12-months
  17 item scale measuring dimensions of emotional adjustments in persons aged 70 to 90. It provides a multidimensional approach to assessing the state of psychological wellbeing and perceived morale using three factors: agitation, attitude toward own aging and lonely satisfaction. Total score ranges from 0-17 with higher scores indicating higher morality.
The NIH Toolbox Meaning and Purpose Short Form | 4-months
  8-item, form that assesses the degree to which participants feel their lives matter/make sense. Each item is rated on a 5-point Likert scale with responses ranging from "strongly disagree" to "strongly agree" and from "not at all" to "very much." Total score ranges from 8-40 with higher scores indicating better outcomes.
The NIH Toolbox Meaning and Purpose Short Form | 8-months
  8-item, form that assesses the degree to which participants feel their lives matter/make sense. Each item is rated on a 5-point Likert scale with responses ranging from "strongly disagree" to "strongly agree" and from "not at all" to "very much." Total score ranges from 8-40 with higher scores indicating better outcomes.
The NIH Toolbox Meaning and Purpose Short Form | 12-months
  8-item, form that assesses the degree to which participants feel their lives matter/make sense. Each item is rated on a 5-point Likert scale with responses ranging from "strongly disagree" to "strongly agree" and from "not at all" to "very much." Total score ranges from 8-40 with higher scores indicating better outcomes.
The Patient Health Questionnaire-9 (PHQ-9) | 4-months
  Reliable and valid (in a variety of patient populations) multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. Response options are provided on a 4-point Likert scale, with total score ranging from 1-27. Lower scores indicate better outcomes.
The Patient Health Questionnaire-9 (PHQ-9) | 8-months
  Reliable and valid (in a variety of patient populations) multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. Response options are provided on a 4-point Likert scale, with total score ranging from 1-27. Lower scores indicate better outcomes.
The Patient Health Questionnaire-9 (PHQ-9) | 12-months
  Reliable and valid (in a variety of patient populations) multipurpose instrument for screening, diagnosing, monitoring, and measuring the severity of depression. Response options are provided on a 4-point Likert scale, with total score ranging from 1-27. Lower scores indicate better outcomes.
The Center for Epidemiological Studies-Depression (CES-D) | 4-months
  20-item measure that rates how often over the past week respondents have experienced depressive symptoms. Response options are provided on a 4-point Likert scale with total scores ranging from 0-60. Lower scores indicate lower depressive symptoms.
The Center for Epidemiological Studies-Depression (CES-D) | 8-months
  20-item measure that rates how often over the past week respondents have experienced depressive symptoms. Response options are provided on a 4-point Likert scale with total scores ranging from 0-60. Lower scores indicate lower depressive symptoms.
The Center for Epidemiological Studies-Depression (CES-D) | 12-months
  20-item measure that rates how often over the past week respondents have experienced depressive symptoms. Response options are provided on a 4-point Likert scale with total scores ranging from 0-60. Lower scores indicate lower depressive symptoms.
The State-Trait Anxiety Inventory (STAI) | 4-months
  Commonly used measure of anxiety with 40 total items. Response options are provided on a 4-point Likert scale. Total score range from 40-160 with lower scores indicating lower anxiety.
The State-Trait Anxiety Inventory (STAI) | 8-months
  Commonly used measure of anxiety with 40 total items. Response options are provided on a 4-point Likert scale. Total score range from 40-160 with lower scores indicating lower anxiety.
The State-Trait Anxiety Inventory (STAI) | 12-months
  Commonly used measure of anxiety with 40 total items. Response options are provided on a 4-point Likert scale. Total score range from 40-160 with lower scores indicating lower anxiety.
The General Self-Efficacy Scale (GSE) | 4-months
  10-item psychometric scale that assesses optimistic self-beliefs to cope with a variety of difficult demands in life. Response options are provided on a 4-point Likert scale with total score ranging from 10-40. Higher total score indicates better outcomes.
The General Self-Efficacy Scale (GSE) | 8-months
  10-item psychometric scale that assesses optimistic self-beliefs to cope with a variety of difficult demands in life. Response options are provided on a 4-point Likert scale with total score ranging from 10-40. Higher total score indicates better outcomes.
The General Self-Efficacy Scale (GSE) | 12-months
  10-item psychometric scale that assesses optimistic self-beliefs to cope with a variety of difficult demands in life. Response options are provided on a 4-point Likert scale with total score ranging from 10-40. Higher total score indicates better outcomes.
Multifactorial Memory Questionnaire (MMQ) | 4-months
  A measure constructed to reflect aspects of memory that are potentially amenable to clinical intervention. The Contentment subscale contains 18 statements that assess emotions and perceptions about current memory ability including anxiety, embarrassment, and irritability. The Ability subscale contains 20 items phrased as memory failures in everyday memory situations (e.g., forgetting an appointment). The Strategy subscale measures self-reported cognitive strategy use. Response options are provided on a 5-point Likert scale. Total score ranges from 0-80 with higher scores indicating better outcomes.
Multifactorial Memory Questionnaire (MMQ) | 8-months
  A measure constructed to reflect aspects of memory that are potentially amenable to clinical intervention. The Contentment subscale contains 18 statements that assess emotions and perceptions about current memory ability including anxiety, embarrassment, and irritability. The Ability subscale contains 20 items phrased as memory failures in everyday memory situations (e.g., forgetting an appointment). The Strategy subscale measures self-reported cognitive strategy use. Response options are provided on a 5-point Likert scale. Total score ranges from 0-80 with higher scores indicating better outcomes.
Multifactorial Memory Questionnaire (MMQ) | 12-months
  A measure constructed to reflect aspects of memory that are potentially amenable to clinical intervention. The Contentment subscale contains 18 statements that assess emotions and perceptions about current memory ability including anxiety, embarrassment, and irritability. The Ability subscale contains 20 items phrased as memory failures in everyday memory situations (e.g., forgetting an appointment). The Strategy subscale measures self-reported cognitive strategy use. Response options are provided on a 5-point Likert scale. Total score ranges from 0-80 with higher scores indicating better outcomes.
The Montreal Cognitive Assessment (MoCA) | 4-months
  Screening instrument that assesses multiple cognitive domains with total score ranging from 0 to 30 points, and a cut score of 24 has demonstrated very good specificity (by correctly identifying 87% of healthy participants) and excellent sensitivity when differentiating MCI (90%) and Alzheimer disease (100%) from healthy comparisons. Total score ranges from 0-30 with higher score indicating better outcomes.
The Montreal Cognitive Assessment (MoCA) | 8-months
  Screening instrument that assesses multiple cognitive domains with total score ranging from 0 to 30 points, and a cut score of 24 has demonstrated very good specificity (by correctly identifying 87% of healthy participants) and excellent sensitivity when differentiating MCI (90%) and Alzheimer disease (100%) from healthy comparisons. Total score ranges from 0-30 with higher score indicating better outcomes.
The Montreal Cognitive Assessment (MoCA) | 12-months
  Screening instrument that assesses multiple cognitive domains with total score ranging from 0 to 30 points, and a cut score of 24 has demonstrated very good specificity (by correctly identifying 87% of healthy participants) and excellent sensitivity when differentiating MCI (90%) and Alzheimer disease (100%) from healthy comparisons. Total score ranges from 0-30 with higher score indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen O'Connor, PsyD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (1):
- VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No